CLINICAL TRIAL: NCT00818675
Title: A Randomized Discontinuation Phase II Trial of Ridaforolimus in Non-Small Cell Lung Cancer (NSCLC) Patients With KRAS Mutations
Brief Title: A Study of Ridaforolimus in Non-Small Cell Lung Cancer (NSCLC) Patients With Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Mutations (MK-8669-021 AM1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8669-021; 2008_599
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ridaforolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ridaforolimus (Experimental)
  Interventions: Drug: Lead-In Ridaforolimus; Drug: Comparator: Blinded Ridaforolimus
- Placebo (Placebo Comparator)
  Interventions: Drug: Lead-In Ridaforolimus; Drug: Comparator: Blinded Placebo

INTERVENTIONS:
Drug: Lead-In Ridaforolimus — Four 10mg tablets of ridaforolimus once daily for five consecutive days each week followed by 2 days days of treatment holiday, during the 8 week lead in treatment period.
  Other Names: MK-8669; AP23573; Deforolimus (until May, 2009)
Drug: Comparator: Blinded Ridaforolimus — Four tablets of blinded ridaforolimus administered daily for 5 consecutive days each week followed by 2 days days of treatment holiday
  Other Names: MK-8669; AP23573; Deforolimus (until May, 2009)
  Arms: Ridaforolimus
Drug: Comparator: Blinded Placebo — Four tablets of blinded placebo (to match ridaforolimus) administered daily for 5 consecutive days each week followed by 2 days of treatment holiday
  Arms: Placebo

SUMMARY:
This is a randomized discontinuation study of ridaforolimus in patients with advanced NSCLC who have failed at least 1 but no more than 3 prior treatment regimens and who have KRAS mutant lung cancer. Following 8 weeks of open-label ridaforolimus lead-in there will be an assessment of disease status. Patients assessed by the investigator to have stable disease after 8 weeks will be randomized to double-blind treatment with ridaforolimus or placebo. Patients assessed to have partial or complete response will continue on open-label ridaforolimus. Patients assessed to have disease progression will be discontinued from study.

DETAILED DESCRIPTION:
Allocation and Arms Additional Information: All Patients will receive an 8-week

open-label lead-in treatment of ridaforolimus. After this 8 week period patients will be re-assessed for disease status. Patients who are stable after 8 weeks are randomized in a double-blind fashion to continue treatment with ridaforolimus or to a placebo until disease progression. (Those patients who have stable disease but are randomized to placebo may cross-over to open-label ridaforolimus at the time of disease progression.)

Those patients with tumor shrinkage during the open-label lead-in treatment will continue on open-label ridaforolimus, while those patients who have disease progression at 8-weeks are taken off-study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically confirmed stage IIIB/IV non-small cell lung cancer
* Patient has a documented mutation of the KRAS gene
* Patient has evidence of disease progression following 1 but no more than 3 prior chemotherapy regimens
* A minimum of 4 weeks has passed since the most recent anti-cancer treatment
* Women of childbearing potential must have a negative pregnancy test prior to start of therapy and must use an approved contraceptive method for the duration of the study
* Patient has adequate organ function
* Patient has performance status of <=2 on Eastern Cooperative Oncology Group (ECOG) performance scale
* Patient is >=18 years of age

Exclusion Criteria:

* Patient has received more than 2 prior chemotherapy regimens for the treatment lung cancer
* Patient is known to have active brain metastases
* Patient is currently participating or has participated in an investigational drug study within 30 days
* Patient is known to be Human Immunodeficiency Virus (HIV) positive or has a known history of Hepatitis B or C
* Patient has an active infection requiring prescribed intervention
* Patient has newly diagnosed or un-controlled Type 1 or 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in the randomized population | Randomization (Week 8) and every 8 weeks until progressive disease or death

SECONDARY OUTCOMES:
Overall response rate (ORR) in the full analysis population | Study entry (Visit 1) and every 8 weeks until progressive disease or death
Overall survival (OS) in the full analysis population | From study entry (Visit 1) to death due to any cause
OS in the randomized population | From study entry (Visit 1) to death due to any cause
PFS in the full analysis population | Study entry (Visit 1) and every 8 weeks until progressive disease or death

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC